CLINICAL TRIAL: NCT03720899
Title: A Pilot Trial Comparing NicoBloc to Nicotine Lozenges: Initial Acceptability and Feasibility Trial
Brief Title: Comparing NicoBloc to Nicotine Lozenges
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karen Cropsey, Professor of Psychiatry, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300001370
Record Dates: First submitted 2018-10-17; First posted 2018-10-25 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Smoking Cessation; Nicotine Dependence
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: participants will be randomized to one of two interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- NicoBloc (Experimental): NicoBloc participants will be provided with NicoBloc to use during counseling sessions and will test smoking their conventional cigarette with NicoBloc.
  Interventions: Drug: NicoBloc
- Nicotine Lozenge (Active Comparator): Participants who receive nicotine lozenge will use the lozenge in session and will discuss the effects of using the lozenge in session.
  Interventions: Drug: Nicotine Lozenge

INTERVENTIONS:
Drug: NicoBloc — For Session 1, participants will use one drop of NicoBloc (which will block 33% of tar and nicotine) on their conventional cigarette and then will smoke this cigarette in session. Following smoking, they will discuss the effects of the NicoBloc on their withdrawal, cravings, and overall enjoyment of their cigarette. To bolster their in vivo NicoBloc experience, participants will be provided with NicoBloc to use between sessions to acclimate to the NicoBloc and to make practice quit attempts (PQAs). Sessions 2 and 3 are similar to Session 1 except they will use more NicoBloc product during the session and will be instructed to use the product between sessions.
  Arms: NicoBloc
Drug: Nicotine Lozenge — Participants who receive nicotine lozenge (mini lozenge) will be given either a 2 or 4 mg lozenge to use in session, depending on how soon they smoke after waking. If a participant smokes within 30 minutes of waking, they start with the 4 mg lozenge; more than 30 minutes, they start with the 2 mg lozenge. They will be given lozenges between sessions to make PQAs.
  Arms: Nicotine Lozenge

SUMMARY:
To examine the feasibility, acceptability, and preliminary impact of using NicoBloc compared to nicotine lozenges

DETAILED DESCRIPTION:
Smoking remains the leading cause of preventable death in the U.S. with approximately 18% of the population continuing to smoke. However, smoking is concentrated in disadvantaged populations where the prevalence of smoking may be as high as 70-80 %. Participants will receive a sampling experience (use of nicotine lozenges or NicoBloc during sessions) with counseling focused around their experience of using these interventions, including side effects and smoking cessation expectancies.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. planning to live in the Birmingham Metro area for the next 3 months
3. Smoking at least 5 cigarettes per day for the past year and a Carbon Monoxide>8ppm to ensure daily smoking. This relatively low cutoff was chosen due to the expectation of enrolling a large >50% African-American average <10 cigarettes per day compared to Whites who average ~15 cigarettes per day
4. exclusive use of filtered cigarettes
5. English speaking.

Exclusion Criteria:

1. Living in a restricted environment that does not allow smoking (e.g., prison or jail facility, etc.)
2. Pregnant or nursing (all women of childbearing potential will be required to use an acceptable form of contraception)
3. Currently enrolled in a smoking cessation treatment program, using nicotine replacement products, or prescribed bupropion or varenicline
4. Known allergy nicotine lozenge
5. Within one month post-myocardial infarction or untreated severe angina
6. Cognitive impairment or unstable psychiatric condition that interferes with the informed consent process (individuals stable on psychiatric medications will be included)
7. Daily or exclusive use of other tobacco products (e.g., electronic cigarettes, little cigars, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Cropsey, Psy.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama, Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Chichester KR, Sisson ML, Chana SM, Wolford-Clevenger C, Hugley MJ, Hawes ES, Palenski P, Nguyen A, Dahne J, Hendricks PS, Cropsey KL. An Open-label Pilot Study of NicoBloc as a Novel Smoking Cessation Intervention. J Addict Med. 2023 Jul-Aug 01;17(4):e269-e277. doi: 10.1097/ADM.0000000000001157. Epub 2023 Mar 3. PMID 37579108

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NicoBloc | Nicotine Lozenge
Started | 21 | 24
Completed | 13 | 13
Not Completed | 8 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NicoBloc | Nicotine Lozenge | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 22 | 40
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 15 | 17 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 17 | 30
  White | 8 | 5 | 13
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: The Treatment Satisfaction Survey
Description: * Number of items: 10
  * Scale: 1 (not at all helpful) - 7 (very helpful), as well as "0" response for "Don't Know".
  * Full-scale range: 0-70
  * Interpretation: Higher scores indicate more treatment satisfaction Subscales: N/A
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NicoBloc | Nicotine Lozenge
Number analyzed (Participants) | 13 | 13
score on a scale | 63.62 (7.04) | 64.67 (17.25)

2. Secondary Outcome: Change in the Questionnaire of Smoking Urges-Brief Form, From Baseline to Week 4 Timepoint
Description: * Number of items: 10
  * Scale: 1 (Strongly Disagree) - 7 (Strongly Agree)
  * Full-scale range: 10-70
  * Interpretation: Higher scores indicate more smoking urges Subscales: N/A
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: Pre - Post Mean Score
Arm/Group | NicoBloc | Nicotine Lozenge
Number analyzed (Participants) | 16 | 17
Pre - Post Mean Score | -1.75 (5.6) | -.65 (5.06)

3. Secondary Outcome: Retention Rates
Description: The total number of participants retained throughout the entirety of the study duration.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | NicoBloc | Nicotine Lozenge
Number analyzed (Participants) | 21 | 24
Participants | 13 | 13

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | NicoBloc | Nicotine Lozenge
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT03720899/Prot_003.pdf
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT03720899/SAP_004.pdf
  • Informed Consent Form (2019-12-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT03720899/ICF_005.pdf